CLINICAL TRIAL: NCT05970653
Title: Effect of Remote Ischemic Conditioning on Cerebral Autoregulation in Patients Undergoing Cerebrovascular Stent Implantation
Brief Title: Effect of RIC on Cerebral Autoregulation in Patients Undergoing Cerebrovascular Stent Implantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of The First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RICCA-CSI
Record Dates: First submitted 2023-07-25; First posted 2023-08-01 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Remote Ischemic Conditioning
Keywords: Remote Ischemic Conditioning; Cerebrovascular Stent Implantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC Group (Active Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg. RIC will be conducted twice daily for 7 consecutive days or from enrollment to discharge.
  Interventions: Procedure: Remote ischemic conditioning
- Sham-RIC Group (Placebo Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg. RIC will be conducted twice daily for 7 consecutive days or from enrollment to discharge.
  Interventions: Procedure: Sham remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg.
  Arms: RIC Group
Procedure: Sham remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg.
  Arms: Sham-RIC Group

SUMMARY:
The purpose of this study is to determine the effect of remote ischemic conditioning on cerebral autoregulation in patients undergoing cerebrovascular stent implantation.

DETAILED DESCRIPTION:
In this study, 104 cases of patients with cerebrovascular stent implantation will be enrolled in the First Hospital of Jilin University, and they will be divided into the RIC group and the sham-RIC group. The RIC group received remote ischemic conditioning for 200mmHg, 2 times per day for 7 consecutive days or from enrollment to discharge. The sham-RIC group received remote ischemic conditioning for 60mmHg, 2 times per day for 7 consecutive days or from enrollment to discharge. Two groups will be followed up to evaluate the effect of remote ischemic conditioning on cerebral autoregulation in patients undergoing cerebrovascular stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years, regardless of sex;
* Patients with symptomatic or asymptomatic cerebral vascular stenosis (including internal carotid artery system and vertebrobasilar system) who are candidates for elective cerebrovascular stenting.
* Patients or their immediate family members are able and willing to sign informed consent.

Exclusion Criteria:

* Patients with progressive stroke;
* mRS≥ 2 points before admission;
* Patients with other surgical treatments;
* Patients with other serious diseases or a life expectancy of less than 3 months
* Patients who had contraindication of remote ischemic conditioning, such as severe soft tissue injury, fracture or vascular injury in the upper extremities, venous thrombosis in the acute or subacute stage of upper extremities;
* Laboratory test indicators are unqualified: aspartate aminotransferase or alanine aminotransferase is 3 times higher than the upper limit of the normal range, blood creatinine > 265umol/L (>3mg/dl), platelet < 100×109/L, international normalized ratio (INR), activated partial thromboplastin time (APTT), prothrombin time (PT) exceed the upper limit of the normal range;
* Pregnant or lactating women;
* Patients who are participating in other clinical studies, or who have participated in other clinical studies within 3 months prior to enrollment;
* Unwillingness to be followed up or poor adherence to treatment;
* Other circumstances that the investigator considers unsuitable for enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral autoregulation parameter | 0-7 days
  Cerebral autoregulation parameters derived from transfer function analysis. Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the autoregulatory parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China